CLINICAL TRIAL: NCT06569589
Title: Tissue Sodium Quantification in Patients With Primary Aldosteronism
Brief Title: Tissue Sodium Quantification in Patients With Primary Aldosteronism: See Sodium to Treat
Acronym: SSTT
Status: Recruiting | Type: Observational
Sponsor: Jens Titze (Other)
Collaborators: Changi General Hospital (Other); Singapore General Hospital (Other); Sengkang General Hospital (Other)
Responsible Party: Sponsor-Investigator, Jens Titze, Associate Professor, Duke-NUS Graduate Medical School
Organization: Duke-NUS Graduate Medical School (Other)
Other Study IDs: 2023-1047
Record Dates: First submitted 2024-08-01; First posted 2024-08-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Primary Aldosteronism; Hypokalemia
Keywords: NaMRI; muscle Na+ quantification; K+ supplementation
MeSH Terms: conditions — Hypertension; Hyperaldosteronism; Hypokalemia | interventions — Potassium, Dietary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Suspected PA: Age 21-70 years, with arterial hypertension or suspected to have primary aldosteronism based on Endocrine Society Guidelines.
  Interventions: Diagnostic Test: 23NaMRI Scan; Dietary Supplement: Potassium Chloride (KCl)

INTERVENTIONS:
Diagnostic Test: 23NaMRI Scan — 23NaMRI, a non-invasive detection and quantification of hidden tissue Na+ stores in humans.
Dietary Supplement: Potassium Chloride (KCl) — K+ supplementation intervention is given participants as part of their standard care. In this trial the K+ supplementation dosage is standardized and adjusted based on blood K+ level

SUMMARY:
The study aims to provide quantitative facts on the pathophysiological changes in tissue Na+ content during Na+/K+ redistribution disorders in patients with PA in response to standard therapy. The investigators hypothesize that patients with primary aldosteronism have excessive Na+ storage in the muscle, which can now be quantified non-invasively using 23NaMRI. In analogy to the role of HbA1c as a metabolic long-term marker in diabetes, the quantifiable changes in muscle Na+ content may deliver the data evidence necessary to justify and conduct randomized diagnostic endpoint outcome trials in the future, with the ultimate aim to improve PA detection rate and treatment.

DETAILED DESCRIPTION:
Arterial hypertension is a major modifiable cardiovascular risk factor along with diabetes mellitus. Hypertension due to autonomous elevation in aldosterone production (Primary Aldosteronism; PA) is not responsive to usual antihypertensive medications and is dramatically underdiagnosed in standard clinical routine. Currently, only 0.1% (1,280,000 worldwide and 1,140 Singaporeans) are diagnosed, much lower than the 5-20% (64,000,000-256,000,000 worldwide and 57,000-228,000 Singaporeans) of all patients with arterial hypertension estimated to suffer from PA. Given the high prevalence of PA, low rates of diagnoses, high cardiometabolic morbidity and mortality associated with untreated PA, the detection of more patients with PA is obligatory, and treatment success must be monitored.

The investigators hypothesize that patients with primary aldosteronism have excessive Na+ storage in the muscle, which can now be quantified non-invasively using 23NaMRI. This study will be the first to systematically quantify changes in muscle Na+ stores in these patients in response to standard therapy. There is currently no established clinical diagnostic tool to detect or quantify the underlying cellular Na+/K+ redistribution physiology in patients with PA. Seeing and quantifying the Na+ non-invasively with 23NaMRI will provide a fresh "look" into the pathophysiological principles of solute and fluid homeostasis to evaluate therapy efficacy, and to improve rates of PA diagnoses with an intention to cure.

This is a prospective non-randomized multi-centre study with 3 study visits ( pre-potassium treatment, pre- diagnosis and post-treatment) over a study period of 3 years. Approximately 100 participants will be recruited from hospital sites. The purpose of the study is to detect and quantify a hidden pathophysiological Na+/K+ redistribution process at the tissue level, using 23NaMRI, in an effort to provide an alternative to traditional hormone and solute diagnostics in blood and urine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-70 years, with arterial hypertension or suspected to have primary aldosteronism based on Endocrine Society Guidelines.
2. Male and female patients older than 21 years.
3. Willingness to participate and ability to provide informed consent.

Exclusion Criteria:

1. Patients with exclusion criteria for the MRI, such as:

   * implanted devices (surgical clips, heart pacemakers or defibrillators, cochlear implants)
   * iron-based tattoos
   * any other pieces of metal or devices that are not MR-Safe anywhere in the body
   * patients who exhibit noticeable anxiety and/or claustrophobia into the MRI scanner
   * pregnancy
2. Diagnosis of heart failure NYHA classes III and IV
3. Impaired renal function with eGFR<30 ml/min or proteinuria > 1 g/24h
4. Liver disease with cirrhosis (Child-Pugh class C) or hypoalbuminemia
5. Muscular dystrophies
6. Patients with active cancer or severe comorbid conditions likely to compromise survival or study participation
7. Unwillingness or other inability to cooperate

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 patients with hypertension with accompanying hypokalemia will be recruited from hospital sites.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Patients with primary aldosteronism have a 10-20% higher muscle Na+ content compared to healthy controls | Baseline
  Difference in muscle Na+ content as measured with 23NaMRI between patients with PA and healthy controls at baseline.

SECONDARY OUTCOMES:
High K+ intake reduces muscle Na+ in patients with primary aldosteronism | Baseline to 3 Months
  Change in muscle Na+ content as measured with 23NaMRI, 3 months after initiation of K+ supplementation
MR blockade reduces muscle Na+ conten in patients with primary aldosteronism | Baseline to 18 months
  Change in muscle Na+ content as measured with 23NaMRI, 12-18 months after initiation of MR blockade treatment
Compared to MR blockade, adenoma surgical removal is more efficient in reducing muscle Na+ in patients with primary aldosteronism | 36 Months
  Change in muscle Na+ content as measured with 23NaMRI after adenoma surgical removal compared to MR blockade treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Titze, MD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (4):
- Singapore (4):
  - Singapore General Hospital, Singapore
  - Duke NUS Medical School, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during study visits will be shared for participants who have provided informed consent for data sharing
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years after article publication with no end date
Access Criteria: Access will be granted upon reasonable request, provided that interested researchers have a scientific hypothesis for which they submit a methodologically sound proposal, including clearly defined research hypothesis and a statistical analysis plan.

REFERENCES:
- [Background] Kopp C, Linz P, Wachsmuth L, Dahlmann A, Horbach T, Schofl C, Renz W, Santoro D, Niendorf T, Muller DN, Neininger M, Cavallaro A, Eckardt KU, Schmieder RE, Luft FC, Uder M, Titze J. (23)Na magnetic resonance imaging of tissue sodium. Hypertension. 2012 Jan;59(1):167-72. doi: 10.1161/HYPERTENSIONAHA.111.183517. Epub 2011 Dec 5. PMID 22146510
- [Background] Kopp C, Linz P, Dahlmann A, Hammon M, Jantsch J, Muller DN, Schmieder RE, Cavallaro A, Eckardt KU, Uder M, Luft FC, Titze J. 23Na magnetic resonance imaging-determined tissue sodium in healthy subjects and hypertensive patients. Hypertension. 2013 Mar;61(3):635-40. doi: 10.1161/HYPERTENSIONAHA.111.00566. Epub 2013 Jan 21. PMID 23339169
- [Background] Marton A, Saffari SE, Rauh M, Sun RN, Nagel AM, Linz P, Lim TT, Takase-Minegishi K, Pajarillaga A, Saw S, Morisawa N, Yam WK, Minegishi S, Totman JJ, Teo S, Teo LLY, Ng CT, Kitada K, Wild J, Kovalik JP, Luft FC, Greasley PJ, Chin CWL, Sim DKL, Titze J. Water Conservation Overrides Osmotic Diuresis During SGLT2 Inhibition in Patients With Heart Failure. J Am Coll Cardiol. 2024 Apr 16;83(15):1386-1398. doi: 10.1016/j.jacc.2024.02.020. PMID 38599715